CLINICAL TRIAL: NCT03475043
Title: Neuroplasticity in Auditory Aging_Auditory Temporal processing_Project 2
Brief Title: Neuroplasticity in Auditory Aging_Project 2 Aims 1 and 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Sandra Gordon Salant, Professor, University of Maryland, College Park
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UMDCP_P01P2; P01AG055365 (NIH)
Record Dates: First submitted 2018-03-15; First posted 2018-03-23 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Auditory Perceptual Disorders; Aging Problems
MeSH Terms: conditions — Auditory Perceptual Disorders

STUDY DESIGN:
Intervention Model Description: Experimental group Active control group Passive control group
Who Masked: Outcomes Assessor
Masking Description: Examiners who conduct pre, post, and retention tests with participants do not know to which group a participant is assigned (experimental group, active control group, passive control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Auditory training: temporal cues (Experimental): Aim 1: Listeners will hear target acoustic stimuli that vary in a temporal (timing/duration) cue for 9, 1-hour training sessions and will receive correct-answer feedback.
  Aim 2: Listeners will hear sentences that vary in speech rate for 6, 1-hour training sessions and will receive correct-answer feedback.
  Interventions: Behavioral: Auditory training: temporal cues
- Auditory training: non-temporal cues (Active Comparator): Aim 1: Listeners will hear target acoustic stimuli that vary in either stimulus intensity or stimulus frequency during 9, 1-hour training sessions and will receive correct-answer feedback.
  Aim 2: Listeners will hear speech in varying levels of noise during 6, 1-hour training sessions and will receive correct-answer feedback.
  Interventions: Behavioral: Auditory training: temporal cues
- Passive control group (Aims 1 and 2) (No Intervention): Listeners will be evaluated on pre-training and post-training tests, but will receive no training at all.

INTERVENTIONS:
Behavioral: Auditory training: temporal cues — Behavioral training for 6-9 hours in listening to specific characteristics of acoustic signals. Listeners receive correct-answer feedback on each trial.
  Other Names: Auditory training: non-temporal cues
  Arms: Auditory training: non-temporal cues; Auditory training: temporal cues

SUMMARY:
Millions of elderly adults in the USA have age related hearing loss (ARHL), a malady that affects half of adults 60-69 years, and the majority of older adults. This hearing loss not only impacts communication and functional ability, but also is strongly associated with cognitive decline and decreased quality of life. This project aims to develop effective strategies to compensate and reverse this process through a deeper understanding of plasticity and adaptive auditory function, and how to engage it and harness it to remedy ARHL.

DETAILED DESCRIPTION:
The detrimental effects of aging on auditory temporal processing have been well documented in humans and animal models. At present, there are gaps in knowledge of the extent to which these auditory temporal processing deficits can be mitigated in older adults with or without hearing loss through auditory training and neuroplasticity, to improve precision of neural timing and speech understanding. The long-term goal is to determine the extent to which hearing deficits in older adults can be ameliorated with auditory training. The investigators propose an innovative approach to the investigation of aging, hearing, and neuroplasticity by marrying perceptual training experiments with electrophysiological measurements. The objectives are to compare young normal-hearing (YNH), older normal-hearing (ONH), and older hearing-impaired (OHI) adult listeners, and evaluate the improvements in perceptual and electrophysiological measures of temporal processing after explicit training on auditory temporal processing tasks. The central hypothesis is that training of auditory temporal processing will produce concomitant improvements in both perceptual performance and neural encoding, which will close the gap in the age-related differences between groups. The central hypothesis will be tested by pursuing two specific aims: (Aim 1) Determine the extent to which perceptual training on temporal rate discrimination using simple non-speech stimuli improves perceptual and neural encoding in YNH, ONH, and OHI listeners; and (Aim 2) Determine the extent to which perceptual training on the processing of sentences with increasing presentation rate can improve behavioral performance and neural encoding in YNH, ONH, and OHI listeners. The expected outcomes are that the investigators will learn what perceptual training tasks lead to simultaneous improvements in perceptual and neural auditory temporal processing and the findings will produce a significant impact in older listeners who experience difficulty in communicating in daily life because they will lead directly to focused and novel forms of rehabilitation. This research is innovative because the investigators will have established techniques that are proven to provide significant improvements in auditory temporal processing and speech perception, combined with evidence of improvements to neural encoding. These studies will serve the larger goals of the program project grant because they will help identify the neuroplastic mechanisms in the brain of humans that correspond to successful behavioral outcomes in younger and older adults.

ELIGIBILITY:
Inclusion Criteria:

* native speaker of English
* normal cognitive function as measured on Montreal Cognitive Assessment
* pass screening auditory brainstem response test to make sure they have recordable brainwaves to acoustic stimuli
* age and hearing sensitivity:
* young normal-hearing listeners, 18-35 years, hearing thresholds less than 25 decibels (dB) HL from 250 - 4000 Hz;
* older normal-hearing listeners, 65-85 years, hearing thresholds less than 25 dB HL, from 250-4000 Hz;
* older hearing-impaired listeners, 65-85 years, with mild-to-moderate, high frequency sensorineural hearing loss;
* high school diploma

Exclusion Criteria:

* absence of conductive hearing loss and middle-ear disease
* no neurological disease
* severe or profound hearing loss
* non-native speaker of English
* cognitive impairment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Improvement in behavioral auditory temporal processing measures (Aim 1) | completion of study, approximately 30 months
  Decrease in threshold (in msec) for discriminating a comparison pulse train to a standard, decrease in cross-over points (in msec) for trained word contrasts, and increase in rate of speech for 50% correct recognition
Improvement in recognition of trained stimuli - fast speech (Aim 2) | completion of study, approximately 24 months
  Increase in speech rate at which listener maintains 50% and 80% correct recognition

SECONDARY OUTCOMES:
Change in spectral energy and neural phase locking for trained stimuli (Aim 1) | completion of study, approximately 30 months
  Increase in spectral energy for pulse trains, cessation of neural phase locking for trained words during silent intervals of the word, and increase in phase-locking factor following training of time-compressed speech, as measured on the Auditory Steady-State Response
Change in phase locking to trained or equivalent stimuli (Aim 2) | completion of study in approximately 24 months
  Increase in phase-locking factor following training of time-compressed speech, as measured in the frequency-following response
Change in reconstruction accuracy to trained or equivalent stimuli (Aim 2) | completion of study in approximately 24 months
  Increase in reconstruction accuracy following training of time-compressed speech, as measured with envelope tracking to five-minute speech samples

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Gordon-Salant, Ph.D., Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, College Park, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share the final dataset that includes initial assessment information, behavioral performance pre-training and post-training data, and neurophysiologic data. Any shared dataset(s) will be stripped of protected health information (PHI) before release, and the investigators will make the data and associated documentation available only to IRB-approved colleagues and collaborators under an agreement that provides for: (1) a commitment to using the data only for research purposes and not to inappropriately identify any individual participant; and (2) a commitment to securing the data using appropriate information technology and practices.
Supporting Information: Study Protocol
Time Frame: Six months after publication until May 31, 2022
Access Criteria: The data will be available only to Institutional Review Board-approved colleagues and collaborators under an agreement that provides for: (1) a commitment to using the data only for research purposes and not to inappropriately identify any individual participant; and (2) a commitment to securing the data using appropriate information technology and practices. The PI (Gordon-Salant) and co-PI (Anderson) will review requests for access to the data. Once approved, access will be provided by Prometheus Software, LLC. Prometheus will develop best practices for securely sharing research data with our collaborators and the wider scientific community. Finally, Prometheus will ensure that the project complies with all relevant data distribution agreements and data submission requirements.